CLINICAL TRIAL: NCT05800522
Title: A Randomized Controlled Effectiveness Trial of a Transdiagnostic Parent Training Intervention to Prevent Childhood Mental Health Problems in Norwegian Frontline Services
Brief Title: Testing the Effectiveness of Supportive Parents - Coping Kids
Acronym: SPARCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Child Behavioral Development (Other)
Collaborators: Kavli Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 50708
Record Dates: First submitted 2023-02-28; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-02

CONDITIONS: Conduct Problems; Anxiety Symptoms; Depressive Symptoms
Keywords: Transdiagnostic prevention; Childhood mental health problems; Parent training; Adaptive intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A two-armed parallel randomized effectiveness trial in Norwegian frontline services.
Who Masked: Participant
Masking Description: Participants are to be masked to what treatment condition they are assigned to, whether they receive the treatment or control condition. Treatment conditions are termed group 1 and group 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Various active treatments implemented in Norwegian frontline services. Treatments will include different measures varying in scope and intensity including eclectic counselling and other systematic and evidence-based interventions.
  Interventions: Behavioral: Behavioral parent or child directed intervention
- Intervention group (Experimental): Transdiagnostic and preventive parent training intervention, Supportive parents - coping kids (SPARCK)
  Interventions: Behavioral: Supportive Parents - Coping Kids

INTERVENTIONS:
Behavioral: Behavioral parent or child directed intervention — Control group will include different behavioral interventions that may include caretakers or the target child, and thus may vary in scope and intensity.
  Arms: Control group
Behavioral: Supportive Parents - Coping Kids — Intervention group will receive the transdiagnostic parent intervention (SPARCK). SPARCK is designed to include up to 12 sessions with caretakers. If necessary and applicable, children can attend sessions. The starting point for the development of SPARCK has been the Social Interaction Learning model, which represents the behavioral management perspective. In addition, SPARCK consists of empirically supported components based on attachment theory, emotion socialization, CBT, and family accommodation. Thus, content and strategies have been collected from different theories to provide a diverse toolkit tailored to address transdiagnostic problems in families with externalizing, internalizing, and caregiver challenges. SPARCK content and target strategies are tailored to the needs of the families and children, and the manual explains the content and how the target strategies may be tailored and combined.
  Other Names: Parent training intervention
  Arms: Intervention group

SUMMARY:
The aim of this clinical trial is to test the effectiveness of the parent training intervention Supportive Parents - Coping Kids (SPARCK) for prevention of childhood mental health problems. The main research questions are:

• Is SPARCK effective in preventing and reducing negative outcomes and promoting positive outcomes for eligible children and parents compared with regular care practice?

In addition, investigators will conduct an implementation study to examine relations between implementation determinants and implementation and clinical outcomes in the SPARCK intervention condition

Participants in the effectiveness trial will be randomized to receive either the SPARCK intervention or active regular care practices provided by professionals in the Norwegian frontline services. Researchers will test the effectiveness of the SPARCK intervention at post treatment and six months follow-up.

DETAILED DESCRIPTION:
SPARCK is a novel transdiagnostic and preventive parent intervention targeting parents with children aged 4 to 12 years with elevated, yet subclinical, symptoms of anxiety, depression (internalizing) and/or behavioral problems (externalizing). In this project, investigators will conduct a randomized effectiveness trial with families randomized to SPARCK or regular care practices in the Norwegian frontline services, e.g. child welfare services, health services, and school health services. Investigators will study potential effects of SPARCK primarily on a) child symptoms when compared with regular care, and secondary on b) parenting practices, self-efficacy and stress, c) parent and child stress regulation as indexed by stress hormones (cortisol and DHEA) in hair, d) referrals to specialized services and CWS, and e) child and parent subjective quality of life. Additionally, Investigators will study facilitators and barriers to successful implementation and the relation between implementation and clinical outcomes.

Design: Two-armed parallel group randomized controlled trial. Families will be assessed at three time points: At pre intervention, at post (intervention termination), and at follow-up six months after post assessment. In cases were intervention exceeds 24 weeks, we will assess post at week 25. In such cases, follow-up will be assessed six months after week 25. Stress hormones will be collected at pre intervention and four weeks after intervention termination.

Despite a relatively heterogeneous target group, investigators expect a balanced design in terms of symptom domains and comorbidity across internalizing and externalizing symptoms. However, there is some uncertainty regarding the frequency of children with depressive symptoms exclusively (in contrast to symptoms of anxiety or behavioral problems). Our primary outcomes reflect the transdiagnostic feature of SPARCK; targeting anxiety, depression, and externalizing symptoms. Eligible children may display symptoms symptoms in ether one, two, or across all three symptom domains. Accordingly, investigators do only expect change in a relevant symptom domain if children display elevated levels at pre intervention.

Data will be inspected the data halfway through the data collection to monitor various issues, such as the distribution of symptoms of study families at intake and potential harm to study families. For instance, if children with depressive symptoms exclusively is low-frequent at intake, investigators may modify relevant hypotheses and accompanying primary outcome. An external researcher which is not part of the project will oversee the process.

To investigate the implementation part of the project, investigators will include a quantitative data gathering amongst SPARCK practitioners and their service leaders over three time points; intervention time point 1 (iT1; at project start), iT2 (after one year of data collection), and iT3 (after two years of data collection.).

Recruitment, analysis, and power: Participant recruitment in the effectiveness study will follow regular care procedures for screening and inclusion into the frontline services. Eligible families will be randomized within each site with a 50% chance of being allocated to control or intervention group. To promote predictability for the services in terms of intervention delivery, pairwise randomization within each site will be conducted. To prevent delay of intervention, and if an eligible second case match is not recruited within a four week period, a single block randomization will be done. Blocks are nested within each municipal site and the size of the block is blinded for study personnel and the sites. Randomization will be executed by an external provider, Klinforsk (www.klinforsk.no). The effect of the SPARCK vs. regular care will be indicated through a group (between) by time (within) interaction effect in a mixed effect repeated measures design. With an expected weak effect size of f =0.1, GPOWER 3.1 estimates the necessary n to detect group by time interaction with 80% power to be 164, but this is based on no design effects and no dropout. Assuming a therapist intraclass correlation of 0.08, with 4 cases per therapist, the design effect is 1.24, giving an effective n of 80% of the nominal n. Correcting for design effects and 20 % potential dropout the needed effective sample size is 252.

ELIGIBILITY:
Inclusion Criteria:

* Children displaying elevated symptoms of internalizing or/and externalizing problems

Exclusion Criteria:

* Child is referred to or receives ongoing help in the specialized mental health services for problems in the internalizing or externalizing domains
* Child is diagnosed with psychosis, mental retardation or pervasive developmental disorder
* Acute suicide risk
* Documented or probable ongoing physical or sexual abuse
* Child or caretakers receives other systematic interventions targeting internalizing or externalizing problems while enrolled in the study (prior to 6 month follow-up)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of child anxiety and depression measured by Revised Child Anxiety and Depression Scale | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 47-items instrument tapping children's anxiety and depressive symptoms on a 4-point numeric scale ranging from 1 to 4. A higher score indicates more symptoms
Change in child problem behaviors measured by Eyberg Child Behavior Inventory | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 36-items instrument tapping children's frequency of problem behaviors on a 7 point Likert-scale. Higher scores indicates more problem behavior.

SECONDARY OUTCOMES:
Change in child social and emotional problems measured by the Strengths and difficulties questionnaire (SDQ | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 30-items instrument assessed on a 3-point numeric scale tapping children's internalizing and externalizing problems and prosocial skills. The 20-items total difficulties scale tapping composite internalizing and externalizing symptoms is used as primary outcome measure.
Change in parenting practices measured by Parenting and Family Adjustment Scale (PAFAS) | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 30-items instrument assessed on 4-point Likert scales ranging between "not at all" and "very much" tapping parenting skills and family relationships
Change in parental self-efficacy measured by Me as a Parent (MaaP) | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported short-form 4-item instrument assessed on 5 point Likert scales ranging between strongly disagree and strongly agree tapping parental self-efficacy.
Change in parenting stress measured by the Perceived Stress Scale | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 10-items instrument, assessed on 5-point Likert scales ranging between "never" and "very often ", tapping parents global perception of subjective stress.
Change in stress hormones cortisol and dehydroepiandrosterone (DHEA) | Pre intervention (at respondent study inclusion and post intervention (4 weeks after treatment termination)
  Collected from 2 cm hair samples collected from the primary caretaker and and target-child
Change in parent stress hormones cortisol and dehydroepiandrosterone (DHEA) | Pre intervention (at respondent study inclusion and post intervention (4 weeks after treatment termination)
  Collected from 2 cm hair samples collected from the primary caretaker
Change in child stress hormones cortisol and dehydroepiandrosterone (DHEA) | Pre intervention (at respondent study inclusion and post intervention (4 weeks after treatment termination)
  Collected from 2 cm hair samples collected from the target-child
Change in child subjective quality of life measured by Kid-KINDL | Pre intervention (at respondent study inclusion and post intervention (4 weeks after treatment termination)
  Child reported 24-times instrument, assessed on 5-point Likert scales ranging between "never" and "always", tapping children's perception on quality of life
Prevention of mental health and child protection service use | Two and five years after post intervention (treatment termination)
  Register data on child referrals to specialist mental health services and contact with child protection services retrieved from Norwegian Patient Registry and Statistics Norway, respectively.
Change in parental perceived life quality measured by Satisfaction With Life Scale (SWLS) | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 4-items instrument, assessed on 7-point Likert scales ranging between "strongly disagree" and "strongly agree", tapping parent's global perception of satisfaction with life.
Change in tendency to school refusal measured by SPARCK school refusal scale | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 5-items constructed for the project, assessed on 5-point Likert scales ranging between "very rare" and "very often", tapping child school refusal behavior.

OTHER OUTCOMES:
Feasibility of Intervention Measure (FIM) | Time 1 at project start (March 2023), time 2 after year 1 of data collection (March 2024), and time 3 when data collection is finished (2025))
  Practitioner and service leader reported 4-item scale (Weiner et al., 2017) that measures feasibility of an intervention, which is considered an implementation outcome indicating implementation success. Items are measured on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree).
Acceptability of Intervention Measure (AIM) | Time 1 at project start (March 2023), time 2 after year 1 of data collection (March 2024), and time 3 when data collection is finished (2025)
  Practitioner and service leader reported A 4-item scale (Weiner et al., 2017) that measures acceptability of an intervention, which is considered an implementation outcome indicating implementation success. Items are measured on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness Measure (IAM) | Time 1 at project start (March 2023), time 2 after year 1 of data collection (March 2024), and time 3 when data collection is finished (2025)
  Practitioner and service leader reported 4-item scale that measures appropriateness of an intervention, which is considered an implementation outcome indicating implementation success. Items are measured on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree).
Organizational Readiness for Implementing Change (ORIC) | Time 1 at project start (March 2023), time 2 after year 1 of data collection (March 2024), and time 3 when data collection is finished (2025)
  Practitioner and service leader reported 10-item instrument used to determine a collective level of organizational readiness for change, which is an important factor in successful implementation of new interventions, policies and practices. The measure consists of two subscales labelled Change Commitment (5 items) and Change Efficacy (5 items). Items are measured on a 5-point Likert scale from 1 (Disagree) to 5 (Agree).
Implementation Determinants measure | Time 1 at project start (March 2023), time 2 after year 1 of data collection (March 2024), and time 3 when data collection is finished (2025)
  Practitioner and service leader reported 43-item measure to assess factors that can hinder or foster successful implementation of an intervention into a given context. The measure covers the CFIR domains Innovation (13 items), Outer setting (4 items), Inner setting (7), Individuals (6) and Implementation process (13), which includes several sub-themes/constructs (i.e. innovation relative advantage, innovation complexity, individuals attitudes, skills and motivation, external pressure, tension for change, implementation climate etc.). Items are measured on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree).
SPARCK fidelity measure | Weekly after each SPARCK session during the treatment period (until SPARCK treatment termination)
  SPARCK practitioner reporting intervention content used and client responsiveness
Monitoring of control group intervention content. | Up to three times per case. At treatment start-up and at post treatment (up to 25 weeks). If treatment is not terminated after 25 weeks, at third assessment will be conducted after treatment is terminated.
  Control group practitioner reports of intervention format, content and dosage.
Change in parental psychological distress measured by Hopkins Symptom Checklist (SCL-10) | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 10-items instrument, assessed on 4-point Likert scales ranging between "not at all" and "extremly", tapping parents global perception of psychological distress
Change in family accommodation measured by SPARCK accomodation items | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  14 parent reported items scored on 5-point Likert type scales tapping family accommodation to child problems during the last month.
Changes in child routines measured by SPARCK child routines scale | Pre (at respondent study inclusion), post (at treatment termination or up to 25 weeks), and follow-up (6 months after post assessment)
  Parent reported 3-items, assessed on 5-point Likert scales ranging between "strongly disagree" and "strongly agree", tapping occurrence of morning, meals and bedtime routines, and 4 items on numeric scales ranging between 1 and 4, tapping routine functioning.
SPARCK client satisfaction | Post (at treatment termination or up to 25 weeks)
  Parent reported 5-items constructed for this project, assessed on 5-point Likert scales ranging between "not correct" and "very correct", tapping client satisfaction.
Working Alliance Inventory (WAI) | Post (at treatment termination or up to 25 weeks)
  Parent reported 12-items instrument, assessed on 7-point Likert scales ranging between "never" and "always", tapping parent-client working alliance

CONTACTS AND LOCATIONS:
Overall Officials: Truls Tømmerås, PhD, Principal Investigator — National Center for Child Behavioral Development
Locations (1):
- National Center for Child Behavioral Development, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gronlie AA, Backer-Grondahl A, Nes RB, Gomez MB, Tommeras T. Implementation of a parent training intervention (SPARCK) to prevent childhood mental health problems: study protocol for a pragmatic implementation trial in Norwegian municipalities. Trials. 2024 Dec 21;25(1):846. doi: 10.1186/s13063-024-08704-7. PMID 39709458